CLINICAL TRIAL: NCT01018719
Title: Evaluation of Radiation Induced Cardiotoxicity by Multi-detector Computed Tomography (MDCT)
Brief Title: Evaluation of Radiation Induced Toxicity to the Heart by Multi-detector Computed Tomography (MDCT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Dr. Hadassah Goldberg, Director oncology unit, oncology unit, Western Galilee Hospital, Nahariya, Israel
Other Study IDs: cardiotoxicity66809
Record Dates: First submitted 2009-11-17; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: breast cancer radiotherapy cardiotoxicity multidetector CT; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Multidetector Computed Tomography; Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Left side breast cancer
  Interventions: Device: MDCT, ECG, Echocardiography
- Right side breast cancer
  Interventions: Device: MDCT, ECG, Echocardiography

INTERVENTIONS:
Device: MDCT, ECG, Echocardiography — Multi-detector computed tomography to evaluate coronary artery patency; ECG and Echocardiography - to evaluate cardiac function.

SUMMARY:
The current study is aimed to evaluate various imaging methods, including multidetector computed tomography (MDCT) as potential surrogates to assess the degree of damage caused to the heart by radiation therapy to the breast, in breast cancer survivors many years before it becomes clinically apparent.

DETAILED DESCRIPTION:
Early detection and improved treatment approaches following breast cancer (BC) have increased disease specific survival and resulted in increasing cohorts of BC survivors who are prone to develop late complications from treatment, including damage caused by radiation therapy (RT) to the heart. Older RT techniques for treating the breast resulted in excess cardiovascular morbidity and mortality. Improved RT techniques minimize irradiation to the heart. Data from various trials have yielded conflicting results on the extent to which these contemporary techniques have actually decreased cardiotoxicity. Long term follow-up and large cohorts are needed in order to evaluate the risk for cardiotoxicity, when based on its clinical manifestations. The current study is aimed to evaluate various imaging methods as potential surrogates to assess the degree of damage caused to the heart by RT in BC survivors many years before it becomes clinically apparent.This includes Multi-detector computed tomography (MDCT) - based on high resolution computed tomography of the heart following injection of contrast medium which evaluates the degree of stenosis of the coronary arteries.

One hundred patients treated for breast carcinoma, fifty with left breast and fifty with right breast cancer, will be included in the current study and compared for the incidence of cardiac damage. Since the radiation dose to the heart is substantially lower in patients irradiated for right-sided tumors, comparing the incidence of findings indicating cardiac injury in the two groups will define the contribution of RT to these findings. For each patient included in the study, the incidence of cardiovascular disease will be correlated also with the volume of heart irradiated, the radiation dose delivered to that volume, the concomitant administration of cardiotoxic systemic agents, as well as to patient's age when irradiated and risk factors for developing coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed with early breast cancer, histologically proven. Both invasive and non invasive histologies will be included.
2. The study will include patients, who underwent a definitive surgery - either breast conserving or mastectomy - and received radiation therapy to the breast or to the chest wall respectively +/- to lymphatic drainage.
3. No evidence of recurrence of their malignancy or any other malignant disease.
4. Age at diagnosis and radiation to the breast will not exceed 60 years.
5. Signed informed consent by the patient will be mandatory.

Exclusion Criteria:

1. As MDCT requires injection of contrast media, Patients with contra indications for injection of contrast media, due to either a history of allergic reaction or renal insufficiency, will be excluded of the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with breast cancer followed in the oncology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Degree of damage to the coronary arteries as measured by MDCT | 5 to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Hadassah Goldberg, MD, Principal Investigator — Oncology center, Western Galilee Hospital